CLINICAL TRIAL: NCT06768788
Title: Long-term Evaluation of the Effectiveness of an Intervention Program for Physical Education Teachers Aimed At Increasing Adolescents' Motivation and Physical Activity During Leisure Time
Brief Title: Long-term Impact of PE Teacher Interventions on Adolescent Leisure Time Activity and Motivation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Hasso Paap, Junior Research Fellow in Movement Education, University of Tartu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UTartu
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Physical Activity
Keywords: Autonomy support; Competence support; Relatedness support; Basic psychological needs; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Two-month face-to-face and web-based need-supportive intervention program for PE teachers (Trial 1) (Experimental): The main trial phase 1 For the web-based course, we will create video lectures introducing PE teachers' interpersonal behaviours, students' BPN-s, and different motivational regulations in the field of PE to provide a general overview of the SDT postulates. We will also produce short videos on each need-supportive and need-thwarting behaviour, featuring real-life examples of how to increase specific need-supportive behaviours (a total of 9 videos) and how to avoid each specific need-thwarting behaviour (a total of 13 videos), with an approximate duration of 5-8 minutes for each video. In the face-to-face course, PE teachers will also have the opportunity to experience highly need-supportive and highly need-thwarting PE lessons as students, allowing them to reflect on these experiences later.
  Interventions: Behavioral: Face-to-face and web-based need-supportive intervention program based on the main tenets of SDT in the field of PE 1
- Control group - PE teachers who continue teaching with their existing style (Trial 1) (Other): PE teachers continue their regular teaching and the use of their usual teaching methods and behavioral techniques in PE classes.
  Interventions: Behavioral: Face-to-face and web-based need-supportive intervention program based on the main tenets of SDT in the field of PE 1
- Autonomy or competence or relatedness support intervention (Trial 2) (Experimental): The main trial phase 2 PE teachers participate in one of the three one-month face-to-face and web-based autonomy-supportive, competence-supportive, or relatedness-supportive intervention programs.
  Interventions: Behavioral: Face-to-face and web-based need-supportive intervention program based on the main tenets of SDT in the field of PE 2
- Control group - PE teachers who continue teaching with their existing style (Trial 2) (Other): PE teachers continue their regular teaching and the use of their usual teaching methods and behavioral techniques in PE classes.
  Interventions: Behavioral: Face-to-face and web-based need-supportive intervention program based on the main tenets of SDT in the field of PE 2

INTERVENTIONS:
Behavioral: Face-to-face and web-based need-supportive intervention program based on the main tenets of SDT in the field of PE 1 — Intervention: need support, two-month face-to-face and web-based need-supportive intervention program for PE teachers.
  Arms: Control group - PE teachers who continue teaching with their existing style (Trial 1); Two-month face-to-face and web-based need-supportive intervention program for PE teachers (Trial 1)
Behavioral: Face-to-face and web-based need-supportive intervention program based on the main tenets of SDT in the field of PE 2 — Intervention: autonomy or competence or relatedness support, one-month face-to-face and web-based need-supportive intervention program for PE teachers.
  Arms: Autonomy or competence or relatedness support intervention (Trial 2); Control group - PE teachers who continue teaching with their existing style (Trial 2)

SUMMARY:
This project aims to develop a three-month face-to-face and web-based intervention program for physical education (PE) teachers to increase autonomy, competence, and relatedness supportive behaviour toward their students and to avoid the respective need-thwarting behaviours toward their students. The effectiveness of the intervention program is examined at multiple time points during the three-month period. After the intervention program, it is expected that the experimental group students demonstrate significantly higher intrinsic motivation toward physical activity (PA) and are significantly more physically active, as measured by accelerometers, compared to control group students. Additionally, unique effects of autonomy, competence, and relatedness support interventions on students' intrinsic motivation and PA will be investigated. This project provides highly valuable input for PE teacher training to increase students' intrinsic motivation and their overall PA.

DETAILED DESCRIPTION:
Aim of the study

The main objective of the project is to develop and test the main and combined effects of the PE teachers' face-to-face and web-based need-supportive intervention on Grade 6 to 7 adolescents' leisure time PA. The secondary objective of the project is to test the unique effects of interventions focused on support for each psychological need (i.e., autonomy, competence, and relatedness) separately.

Detailed Description

Background

Research has consistently demonstrated that regular PA is associated with several cognitive, psychological, mental, and physical benefits among adolescents (Rodriguez Ayllon et al., 2019). However, PA levels among adolescents are low worldwide (Sluijs et al., 2021) and tend to decrease with age (Farooq et al., 2018). Low PA during childhood and adolescence increases the risk of chronic diseases in adulthood, leading to higher morbidity and lower quality of life (Mavrovouniotis, 2012). Consequently, researchers aim to identify psychological antecedents of PA to inform effective interventions.

PE lessons provide an ideal environment for conveying health-related messages to adolescents (Powell et al., 2016). PE teachers can support students' autonomy, competence, and relatedness, fostering intrinsic motivation in both PE and leisure-time PA. The trans-contextual model of motivation (TCM) has been extensively used to identify PA determinants in these contexts (Hagger et al., 2003). This model integrates self-determination theory (SDT) (Ryan & Deci, 2017), the theory of planned behaviour (Ajzen, 1991), and Vallerand's hierarchical model of motivation (Vallerand, 1997). One core assumption is that psychological experiences in one context (e.g., PE) influence others (e.g., leisure time) (Hagger et al., 2003). Studies indicate that PE teachers significantly impact students' intrinsic motivation (Aibar et al., 2022; Chang et al., 2016; Kalajas-Tilga et al., 2020). Enhancing PE teachers' autonomy-supportive behaviours is crucial (Reeve & Cheon, 2021). Recent research shows that combining web-based and face-to-face interventions effectively improves PE-related outcomes, such as basic psychological needs (BPN) satisfaction and motivation (Tilga et al., 2021).

Few TCM-guided studies have shown changes in students' PA behaviour during leisure time (e.g., Polet et al., 2021; Schneider et al., 2020), and previous autonomy-supportive interventions have been only partially effective (e.g., Rhodes et al., 2021). There is a scarcity of intervention studies supporting a SDT-based multidimensional approach to promote adolescents' PA participation (Ferriz et al., 2021). Recent findings emphasize the importance of providing autonomy, competence, and relatedness support to fully satisfy BPN-s and enhance intrinsic motivation (Ahmadi et al., in press). It is also crucial to avoid need-thwarting behaviours, as these negatively impact adolescents' outcomes (Ahmadi et al., in press; Haerens et al., 2015; Tilga et al., 2020).

In a Delphi study, Ahmadi and colleagues (2023) classified autonomy, competence, and relatedness support and thwarting behaviours, resulting in a taxonomy of 57 teacher motivational behaviours. A shortlist of 22 behaviours was created by selecting those with mean effect ratings greater than +2, categorized as need-supportive and need-thwarting teaching techniques. This classification is the first to systematically compile expert perspectives on motivational teacher behaviours in education. Building on this taxonomy, researchers can test and apply these behaviours in schools. Ferriz and colleagues (2023) adapted these behaviours to the PE context. This project aims to develop and test an intervention program to enhance PE teachers' supportive behaviours and reduce their thwarting behaviours toward students.

To our knowledge, no studies have combined face-to-face and web-based interventions in PE to enhance teachers' need-supportive behaviours while diminishing need-thwarting behaviours, with the goal of increasing students' intrinsic motivation in PE and leisure-time PA.

Participants

For the main trial phase 1, the statistical power analysis revealed that a minimum sample size of 78 students (i.e., n = 39 students allocated to each of the two study groups) would be required to achieve 80% statistical power to detect medium effect sizes when considering three measurements (baseline vs. one-month vs. three-month follow-up) at the within-subject level (correlated at 0.50), with an alpha level of 0.05. However, considering the possible dropout rate of approximately 40% evident in multiple follow-up studies of physical activity (Duda et al., 2014), the investigators aim to recruit 130 students at baseline (i.e., 65 students allocated to each of the two study groups).

For the main trial phase 2, the statistical power analysis revealed that a minimum sample size of 116 students (i.e., n = 29 students allocated to each of the four study groups) would be required to achieve 80% statistical power to detect medium effect sizes when considering three measurements (baseline vs. one-month vs. three-month follow-up) at the within-subject level (correlated at 0.50), with an alpha level of 0.05. However, considering the possible dropout rate of approximately 40% evident in multiple follow-up studies of physical activity (Duda et al., 2014), the investigators aim to recruit 196 students at baseline (i.e., 49 students allocated to each of the four study groups).

Interventions

Combined face-to-face and web-based need-supportive intervention

There will be four types of different intervention programs:

For the main trial phase 1, there will be a combined face-to-face and web-based autonomy, competence, and relatedness need-supportive intervention program with a duration of two months. During these two months, there will be three face-to-face meetings: at the beginning of the course, at the beginning of the fifth week of the course, and at the beginning of the eighth week of the course (each lasting approximately four hours and consisting of lectures and practical activities with discussions).

Additionally, there will be weekly new materials for PE teachers via a web-based learning platform (Moodle) developed for this project. PE teachers will be required to report weekly on how they provide need support to their students and avoid need-thwarting behaviours through the web-based learning platform. Throughout this online course, PE teachers will receive specific materials about all need-supportive behaviours (a total of 9 specific behaviours) and need-thwarting behaviours (a total of 13 specific behaviours) proposed by Ahmadi and colleagues (2023), and adapted for PE by Ferriz and colleagues (2023). This material contains detailed descriptions of each behaviour along with several real-life examples. Additionally, PE teachers will complete a topic-related test at the end of each week in the online environment to confirm their understanding of the material.

For the main trial phase 2, there will be three different courses:

* A combined face-to-face and web-based autonomy need-supportive intervention program with a duration of one month.
* A combined face-to-face and web-based competence need-supportive intervention program with a duration of one month.
* A combined face-to-face and web-based relatedness need-supportive intervention program with a duration of one month.

All these courses will be identical, with the exception that each course focuses on a specific basic psychological need-autonomy, competence, or relatedness. Each course will begin with a face-to-face meeting, which will be the only face-to-face meeting for that course. The content of this face-to-face meeting will be similar to that of the face-to-face meeting experienced in the main trial phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be qualified full-time secondary school PE teachers and their 6th to 7th grade students, without restrictions on their participation in PE classes.

Exclusion Criteria:

* Students who do not participate in PE classes for health reasons.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Adolescents' participation in leisure time moderate-to-vigorous physical activity (MVPA) | Baseline vs. one-month vs. three-month follow-up
  Behavioural Measure: The primary behavioural outcome measure is adolescents' participation in leisure time moderate-to-vigorous physical activity (MVPA), which will be assessed using Actigraph GT3X accelerometers at baseline, one-month follow-up, and three-month follow-up. In the current study, adolescents' MVPA is measured due to its recognized health benefits, such as improved mental health, enhanced cardiorespiratory fitness, and reduced fat gain among adolescents (Grgic et al., 2018). This project focuses on promoting adolescents' MVPA during their leisure time; therefore, accelerometer data collected during the school day will be excluded from the analyses. Additionally, accelerometer diary data will be utilized to identify the duration of MVPA in both in-school and out-of-school contexts.
Adolescents' Psychological Measures | Baseline vs. one-month vs. three-month follow-up
  Psychological Measures: The self-reported questionnaire includes variables from the trans-contextual model of motivation, such as perceptions of (de-)motivating teaching, assessed using the Situations in School Questionnaire (SIS; Aelterman et al., 2019), adapted to the physical education (PE) context (Diloy-Peña et al., 2023). It will also assess psychological need satisfaction and frustration in PE (Haerens et al., 2015), different forms of motivation in PE (Goudas et al., 1994), and various forms of motivation in the leisure time physical activity context (Ryan & Connell, 1989). Additionally, it will measure attitudes, subjective norms, perceived behavioural control, and intentions for leisure time physical activity (Ajzen, 2003), as well as self-reported physical activity (Godin & Shephard, 1985). Previous research has supported the validity of these measures in an Estonian adolescent sample (Kalajas-Tilga et al., 2022).
PE Teacher Level Measures | Baseline vs. one-month vs. three-month follow-up
  The PE teachers' questionnaire includes self-reported measures of (de-)motivating teaching, assessed using the Situations in School Questionnaire (SIS; Aelterman et al., 2019), adapted to the physical education (PE) context (Diloy-Peña et al., 2023).

CONTACTS AND LOCATIONS:
Overall Officials: Henri Tilga, PhD, Principal Investigator — University of Tartu
Locations (1):
- Institute of Sport Sciences and Physiotherapy, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tilga H, Kalajas-Tilga H, Hein V, Koka A. Web-Based and Face-To-Face Autonomy-Supportive Intervention for Physical Education Teachers and Students' Experiences. J Sports Sci Med. 2021 Oct 1;20(4):672-683. doi: 10.52082/jssm.2021.672. eCollection 2021 Dec. PMID 35321125
- [Background] Kalajas-Tilga H, Koka A, Hein V, Tilga H, Raudsepp L. Motivational processes in physical education and objectively measured physical activity among adolescents. J Sport Health Sci. 2020 Sep;9(5):462-471. doi: 10.1016/j.jshs.2019.06.001. Epub 2019 Jun 8. PMID 32928449
- [Background] Ferriz Morell, R. F., González-Cutre Coll, D., Julián Clemente, J. A. Propuestas didácticas para mejorar la motivación en Educación Física y desarrollar estilos de vida saludable. Barcelona: Inde; 2023.
- [Background] Ahmadi, A., Noetel, M., Parker, P., Ryan, R. M., Ntoumanis, N., et al. A classification system for teachers' motivational behaviors recommended in self-determination theory interventions. Journal of Educational Psychology 2023. DOI: 10.1037/edu0000783